



Centre for Ocular Research & Education (CORE)
School of Optometry & Vision Science | University of Waterloo, 200 University Avenue West | Waterloo, ON, Canada N2L 3G1
+1 519 888-4742 | CORE.uwaterloo.ca

CooperVision, Inc.

EX-MKTG-114

20 May 2020

1.3

### **Protocol**

**Sponsor Company:** 

**Version Number:** 

**Document Date:** 

**Sponsor Study number:** 

**CORE** protocol number:

## COMPARING THE PERFORMANCE OF TWO DIFFERENT DAILY DISPOSABLE LENSES (MIKI)

| Document Type: | Study protocol | |
|---|---|---|
| Clinical Site: | inical Site: CORE, University of Waterloo | |
| This protocol remains the exclusive pro | operty of CORE until it is commissioned by the | e sponsor. |
| Role & printed name | Reviewed and approved (sign) | Date<br>DD/MMM/YYYY |
| Principal investigator: Lyndon Jones | | |
| Lead investigator: Amir Moezzi | | |
| Protocol author: Amir Moezzi | | |
| Quality assurance: Jill Woods | | |
| Sponsor: Jose Vega | | |

#### **Study Personnel**



#### **DOCUMENT CHANGE HISTORY**

| Version # | Author | Description of change(s) | Date |
|---|---|---|---|
| - | | | |
| 1.3 | Amir Moezzi | Revised title; minor wording changes for aligning with the sponsor's preferred formatting | 20may2020 |

#### **Table of contents**

| Do | cument c | change history | 3 |
|----|----------|----------------------------------|----|
| 1 | Introdu | oction | 8 |
| 2 | Objecti | ives | 8 |
| 3 | Hypoth | nesis | 9 |
| 4 | Materia | als and methods | 9 |
| | 4.1.1 | Study design | 9 |
| | 4.1.2 | Overall design | 9 |
| | 4.1.3 | Randomization | 11 |
| | 4.1.4 | Masking | 11 |
| 5 | Study p | population | 11 |
| | 5.1.1 | Sample size calculation | 11 |
| | 5.1.2 | Number of participants | 12 |
| | 5.1.3 | Inclusion and exclusion criteria | 12 |
| | 5.1.4 | Repeated screenings | 13 |
| 5 | 5.2 Stu | udy materials | 13 |
| | 5.2.1 | Lenses | 13 |
| | 5.2.2 | Rewetting drops | 14 |
| | 5.2.3 | Ordering consumables | 14 |
| | 5.2.4 | Contact lens dispensing | 14 |
| | 5.2.5 | Contact lens disposal | 14 |
| | 5.2.6 | Product accountability | 15 |
| 5 | 5.3 Sch | heduled and unscheduled visits | 15 |

| | 5.3 | 3.1 | Study visits | 15 |
|----|------|---------|---------------------------------------------|----|
| | 5.3 | 3.2 | Screening (Visit 1) | 16 |
| | 5.3 | 3.3 | Dispensing lens type #1 (Visit 2) | 17 |
| | 5.3 | 3.4 | 1-week follow-up of lens type #1 (Visit 3) | 19 |
| | 5.3 | 5.5 | Dispensing lens type #2 (Visit 4) | 20 |
| | 5.3 | 5.6 | 1-week follow-up of lens type #2 (Visit 5) | 21 |
| | 5.3 | 5.7 | Study exit | 22 |
| | 5.3 | 8.8 | Unscheduled visits | 22 |
| į | 5.4 | Stu | dy procedures | 22 |
| Ę | 5.5 | | | 23 |
| 6 | Мо | nitor | ing protocol adherence | 23 |
| 7 | Pot | tenti | al risks and benefits to human participants | 24 |
| 8 | Adv | vers | e events | 24 |
| 8 | 3.1 | No | rmal or adaptive symptoms | 26 |
| 8 | 3.2 | Pro | ocedures for adverse events | 27 |
| 8 | 3.3 | Re | porting adverse events | 27 |
| 9 | Dis | cont | tinuation from the study | 28 |
| 10 | De | vice | malfunctions | 29 |
| 11 | Stu | ıdy c | completion and remuneration | 29 |
| 12 | Sta | atistic | cal analysis and data management | 30 |
| , | 12.1 | S | Statistical analysis | 30 |
| , | 12.2 | | Data management | 31 |
| | 12.3 | C | Comments on source documents | 31 |

| 13 | Proto | col training | 31 |
|----|-------|-------------------------------------------------|----|
| 14 | Study | y monitoring | 31 |
| 15 | Study | y management | 32 |
| | 15.1 | Statement of compliance | 32 |
| | 15.2 | Ethics review | 32 |
| | 15.3 | Clinical trial registration | 32 |
| | 15.4 | Protocol deviations | 32 |
| | 15.4. | 1 Major protocol deviations | 33 |
| | 15.4. | 2 Minor protocol deviations | 33 |
| | 15.4. | 3 Reporting and documenting protocol deviations | 33 |
| | 15.5 | Premature termination of the study | 34 |
| | 15.6 | Study participant records | 34 |
| | 15.7 | Retention of study records and data | 34 |
| 16 | Repo | ort | 34 |
| 17 | Refe | rences | 34 |

#### Confidentiality

This is a private document and the property of the Centre for Ocular Research & Education. It is therefore confidential to the recipient and must not be quoted from or distributed beyond the company to which it is sent without the express written permission of the Director (or her/his designate) of the Centre for Ocular Research & Education. Release of information from this document is governed by the research agreement on file.

#### **Disclaimer**

This study will be conducted for research purposes only and is not intended to be used to support safety and efficacy in a regulatory submission.

#### 1 INTRODUCTION

The 2018 International Contact Lens Prescribing report<sup>1</sup> describes 32% of soft lenses are prescribed on a daily disposable (DD) basis worldwide (27% in US), compared with 13% and 51% on a one-to-two week and monthly replacement schedule, respectively (30% and 41% in US). There has been an upward trend in prescribing daily disposables for several years.<sup>2</sup>

Until recently, DD lenses were mainly available in a hydrogel material. However, in line with the increasing market share of DD lens modality, more and more new silicone hydrogel (SiHy) DD lenses are becoming available. One of these new SiHy DD lenses are Precision1 lenses that has been recently introduced by Alcon.

This study will evaluate the performance of Alcon's Precision1 (CONTROL lens) compared to CooperVision's MyDay (TEST lens). All participants will habitually wear soft contact lenses, but they do not have to habitually wear daily disposable lenses. Participants with a history of wearing one of the study contact lenses are not eligible for this study.

. All lenses used in this study are spherical, silicone hydrogel daily disposables lenses that are approved by Health Canada.

#### **2 OBJECTIVES**

The objective of the study is to evaluate and compare the performance of the study TEST lens to the CONTROL lens, when worn on a daily disposable modality over a period of approximately one week each.

The primary outcome variable of this study is:

Overall lens fit acceptance at the 1-week follow-up visit.

The secondary outcome variables are:

- Centration (optimal, slight decentration, moderate decentration but not encroaching limbus, excessive & occasionally encroaching limbus), collected at dispense & 1-week visit;
- Post-blink movement in primary gaze, mm, collected at dispense & 1-week visit;
- Push-up tightness in primary gaze (0-100), collected at dispense & 1-week visit.



#### 3 HYPOTHESIS

The study hypothesis is that:

The study test lens will perform as well or better than the control lens for the ratings of overall fit acceptance at the 1-week follow-up visit.

#### 4 MATERIALS AND METHODS

#### 4.1.1 STUDY DESIGN

#### 4.1.2 OVERALL DESIGN

The study is a prospective, double masked (investigator and participant), bilateral, randomized, one week cross-over dispensing study, which evaluates the study test and control lenses.

Participants will be randomized to wear either the test or the control lens first. All lenses will be worn in a daily disposable lens wear modality for one week (-1/+3 days). The study involve up to 5 scheduled visits. The study design is shown in Figure 1.



Figure 1: Study Design, visits 1 & 2 may be on a single day, also visits 3 & 4 may be on a single day.

<u>Visit 1</u>: Includes screening, baseline assessments, fitting of both study lenses.

<u>Visit 2</u>: Dispense lens pair #1 (either test or control lens, randomized).

Visit 3: 1-week follow-up assessment of lens pair #1

<u>Visit 4</u>: Dispense of lens pair #2 (either test or control lens)

<u>Visit 5</u>: 1-week follow-up assessment of lens pair #2 and study exit.

- Participants will complete the following in-office subjective ratings on paper using a numeric rating scale (0 – 10) at visits 3 and 5 for each lens type:
- Lens handling;







#### 4.1.3 RANDOMIZATION

A randomization schedule will be generated using a web-based program: (for example <a href="https://www.randomization.com">www.randomization.com</a>) by CORE's Data management team, and provided to the research assistants for the study. The schedule will determine the order of lens wear for participants in the study. Study investigators will remain masked to the randomization schedule until the study is completed and the database has been locked.

#### 4.1.4 MASKING

Participants will be masked to the lens assignment. Lenses dispensed to participants may be either over-labelled or have part of the label obscured, however the safety information shall be clearly visible. Investigators will be masked as much as possible however it may not be possible to fully mask the investigators, because identifying lens markings may be visible during the biomicroscopy examination.

#### 5 STUDY POPULATION

#### 5.1.1 SAMPLE SIZE CALCULATION

Sample size was calculated using the mean overall fit acceptance from the previous pilot BOXER study

A sample size of 34 is recommended to detect a mean difference between lens Overall fit acceptance of 0.2 units on the 0 to 4 scale using a standard deviation of 0.4 with 80% power and alpha 0.05 in a two-tailed t-test. Therefore, it is recommended that at least 38 subjects are dispensed in the MIKI study, with a target of 34 to complete.

#### 5.1.2 NUMBER OF PARTICIPANTS

Participants will be screened using CORE records and advertising approved by the UW Office of Research Ethics. Approximately 38 participants will be dispensed with study products in the study, with a target of 34 completing the study.

A documented informed consent process will be conducted with all participants prior to their enrolment in the study and prior to any data collection or measurements.

#### 5.1.3 INCLUSION AND EXCLUSION CRITERIA

A person is eligible for inclusion in the study if he/she:

- 1. Is at least 17 years of age and has full legal capacity to volunteer;
- 2. Has read and signed an information consent letter;
- 3. Is willing and able to follow instructions and maintain the appointment schedule;
- 4. Habitually wears soft contact lenses in daily wear, for minimum of 6-months;
- 5. Is correctable to a visual acuity of 20/40 or better (in each eye) with the study lenses;
- 6. Has an astigmatism of ≤ 1.00 D in subjective refraction;
- 7. Can be fit with study contact lenses with a power between -2.00 and -5.00 DS;
- 8. Demonstrates an acceptable fit with the study lenses;
- Habitually wears single vision soft contact lenses for at least 8 hours per day, 5 days a week, and is willing to wear contact lenses for at least 12 hours a day in the study.

A person may be excluded from the study if he/she:

- 1. Is participating in any concurrent clinical or research study;
- Has any known active\* ocular disease and/or infection;
- 3. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable:
- 4. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
- 5. Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
- 6. Is pregnant, lactating or planning a pregnancy at the time of enrolment because the associated hormonal changes cause changes in the tear layer which impact contact lens comfort. Verbal confirmation at the screening visit is sufficient;
- Has undergone refractive error surgery or any intraocular surgery, including cataract surgery;

- 8. Is an employee of the Centre for Ocular Research & Education;
- 9. Has participated in the BOXER or BASSET Study;
- 10. Has any history of wearing one of the study contact lenses;
- 11. Has participated in any clinical trials within a week prior to the study.
- \* For the purposes of this study, active ocular disease is defined as infection or inflammation, which requires therapeutic treatment. Mild (i.e. not considered clinically relevant) lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and dry eye are not considered active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.

#### 5.1.4 REPEATED SCREENINGS

In some circumstances, a repeated screening may need to be scheduled. The maximum total number of screenings permitted will be 3 ie. 2 re-screens. Examples of reasons include, but are not limited to:

- 1. Incomplete information available at time of screening to determine eligibility (e.g. current lens brands worn, history from current eye care practitioner etc.);
- 2. Study procedures unable to be completed in time scheduled for visit;
- Study products not available at the time of the screening visit;
- The short term use of medications (e.g. antibiotics, antihistamines etc.);
- Reassessment of baseline ocular conditions (e.g. corneal and/or conjunctival staining, scars etc.).

#### 5.2 STUDY MATERIALS

#### **5.2.1 LENSES**

All study lenses are approved by Health Canada. They will be worn bilaterally, and on a daily disposable basis, therefore no lens care solution is required.

Test lens Control lens

Manufacturer CooperVision, Inc. Alcon

Material stenfilcon A verofilcon a

HC licence # 91502 101910

Table 1: Lens characteristics & parameter to be used in the study

| Dk/t (barrer/cm) | 100 | 100 |
|---|---|---|
| Water content | 54% | 51% |
| Sphere power (D) | -2.00 to -5.00 (0.25 steps) | -2.00 to -5.00 (0.25 steps) |
| Base curve (mm) | 8.4 | 8.3 |
| Diameter | 14.2 | 14.2 |
| Replacement schedule | Daily disposable | Daily disposable |

#### 5.2.2 REWETTING DROPS

Participants who habitually use rewetting drops will be asked to refrain during the study, unless necessary for continued lens wear. Participants will keep track of rewetting drop usage, and this will be recorded at each visit. Rewetting drops may be used in the event of any clinical observation and/or adverse event noted during the study.

#### 5.2.3 ORDERING CONSUMABLES

All study lenses (test and control) will be provided by CooperVision.

#### 5.2.4 CONTACT LENS DISPENSING

Lenses will be provided to the participant after being transferred, complete with blister pack solution, to a contact lens cup; this will maintain participant masking and aid investigator masking. The use of saline for rinsing the contact lens prior to insertion is permitted if necessary. Saline will not be dispensed during the study.

#### 5.2.5 CONTACT LENS DISPOSAL

Participants will be instructed to dispose of the worn lenses daily, and return any unworn lenses in their packaging at their next study visit. All contact lenses worn to each 1-week follow up visit will be collected and stored at -80C. These collected lenses will be shipped to CooperVision at the end of the study. The lens deposits will be evaluated and analysed for composition and quantity, no genetic assessments will be conducted.

Additionally, worn lenses associated with adverse events shall be retained at CORE and returned to CooperVision if requested to do so. Typical analysis in these cases relates to inspection for damage and/ or bacterial contamination. No genetic assessments will be conducted.

Upon completion of the study, all non-dispensed and the returned unworn lenses will be destroyed, unless otherwise directed by the study Sponsor.

#### 5.2.6 PRODUCT ACCOUNTABILITY

Accountability logs will be kept to include the number of lenses received, dispensed, unused and, if relevant, returned to sponsor. All products dispensed to each participant will be recorded in the study log.

#### 5.3 SCHEDULED AND UNSCHEDULED VISITS

This study has 5 visits. The visits are as follows:

- Visit 1: Screening, baseline assessments, fitting of both study lenses.
- Visit 2: Dispense lens type #1 (normally combined with Visit 1)
- Visit 3: 1-week follow-up assessment of lens type #1 (6 to 10 days after Visit 2), worn lens collection
- Visit 4: Dispense of lens type #2 (normally combined with Visit 3)
- Visit 5: 1-week follow-up assessment of lens type #2 and study exit (6 to 10 days after Visit 4), worn lens collection

A scheduled follow-up visit may only take place when the participant attends wearing the study lenses for 6-8 hours. If this is not the case and the participant is not experiencing any problems with the lenses, the appointment will be rescheduled, ideally within the visit window.

Visits that fall outside of the specified visit windows will be designated as protocol deviations and at the end of the study, the data collected during protocol deviations will be assessed for their suitability to be included in the analysis population.

#### 5.3.1 STUDY VISITS

The summary of visit codes is shown in Table 2.

Table 2: Summary of visit codes

| Visit # | Day/s | Visit code | Visits | Duration<br>(hours) |
|---|---|---|---|---|
| Visit 1 | 0 | V1<br>(V1R1,& V1R2 for re-screening<br>if required) | Screening, baseline & fit of both study lens | 1.25 |
| Visit 2 | 0 | V2 | Dispense lens type #1 | 0.75 |

| Visit # | Day/s | Visit code | Visits | Duration<br>(hours) |
|---|---|---|---|---|
| | 7 ( 1/+2) after | A23 | | |
| Visit 3 | 7 (-1/+3) after<br>V2 | V3 | 1-week follow-up of type #1 | 0.75 |
| Visit 4 | 7 (-1/+3) after<br>V2 | V4 | Dispense lens type #2 | 0.75 |
| Visit 5 | 7 (-1/+3) after<br>V4 | V5 | 1-week follow-up of type #2 | 0.75 |
| Exit Visit | any | any | Study exit | 0.25 |

#### 5.3.2 SCREENING (VISIT 1)

All participants who sign the informed consent letter will be assigned a study ID number. The investigator will determine participant eligibility using the inclusion and exclusion criteria. Ineligible participants will be discontinued from the study. The procedures to be performed are outlined below:

- The participant is expected to attend the screening / baseline visit wearing their habitual contact lenses.
- The participant will be required to read and sign an Informed Consent Form prior to enrollment. When the participant has signed the consent form, the participant will be considered enrolled in the study.
- Participant demographics and medical history (age, sex, medical conditions, medications, allergies).
- 4. Contact lens history (habitual lens information and wearing habits).



- 7. The participant removes their habitual contact lenses.
- 8.



d.

#### 5.3.3 DISPENSING LENS TYPE #1 (VISIT 2)

The procedures to be performed are outlined below:

- 1. The participant will be assigned a randomization ID (by the research assistant) and the first pair (lens pair #1) of contact lenses (either test or control lens) will be selected according to the randomization table.
- 2. Lens pair #1 will be provided to participants in a manner which does not unmask the participant or investigator, as described in Section 5.2.4.
- 3. The participant will insert the lenses.
- 4. The contact lenses will be allowed to settle for 10 minutes.
- 5. The participant will be asked to give subjective binocular ratings for:
- 6. 7. 8. Lens fit will be assessed and graded according to the following grading scales: c. Lens push-up tightness in primary gaze (0 - 100 scale);

  - d. Centration in primary gaze (scale: optimal, slight decentration, moderate decentration but not encroaching limbus, excessive & occasionally encroaching limbus);
  - e. Post-blink movement in primary gaze (mm);
  - f. Overall fit acceptance (0 4 scale, and reason if Grade 2 or less).



| 10. | |
|-------|--------------------------------------------|
| 5.3.4 | 1-WEEK FOLLOW-UP OF LENS TYPE #1 (VISIT 3) |

Participants will be asked to wear lenses for 6 to 8 hours prior to the visit appointment. Participants who attend without lenses in-situ (wearing lenses) for 6 to 8 hours will be rescheduled (unless they report problems when wearing the lenses).

| 1. | |
|----|------------------------------------------------------------------------|
| 2. | |
| 3. | |
| 4. | |
| _ | |
| 5. | Lens fit will then be assessed and graded according to the CVI grading |
| | scales for the following: |
| | a) |

- b)
- c) Lens push-up tightness in primary gaze (0 100 scale);
- d) Centration in primary gaze (scale: optimal, slight decentration, moderate decentration but not encroaching limbus, excessive & occasionally encroaching limbus);
- e) Post-blink movement in primary gaze (mm);
- f) Overall fit acceptance (0 4 scale) and reason if Grade 2 or less).
- 6. Study lens collection at 1-week: investigator will remove study lenses from participant eyes while wearing a pair of disposable non-latex medical grade gloves. The lenses will be rinsed and stored according to sponsor instructions which will be provided at a later date. They will be labeled with study name, participant study ID, eye, visit# and date without any identifying characteristics. They will be stored in a -80 degrees centigrade freezer and shipped to the sponsor when all participants have completed the study.
- 7. Slit lamp biomicroscopy assessments (see 5.3.2 for details).
- 8. There will be a washout of 10 minutes after lens removal if Visit 4 is to be concurrent with this visit.

#### 5.3.5 DISPENSING LENS TYPE #2 (VISIT 4)

- 1. The participant will be assigned the second pair (lens pair #2) of contact lenses (either test or control lens), which will be selected according to the randomization table.
- 2. Lens pair #2 will be provided to participants in a manner, which does not unmask the participant or investigator, as described in Section 5.2.4.
- 3. The participant will insert the lenses.
- 4. The contact lenses will be allowed to settle for 10 minutes.
- 5. The same procedures will be followed as described in Section 5.3.3 DISPENSING LENS PAIR #1 (VISIT 2), points 5 to 11.
- 6. The participant will be reminded to return for Visit 5 (1-week follow-up visit of study lens #2) and instructed to return used lens foils plus all leftover unworn lenses.

Participants will be asked to wear lenses for 6-8 hours prior to the visit. Participants who attend without wearing lenses for 6-8 hours will be rescheduled (unless they report problems when wearing the lenses).

- 1. The same procedures will be carried out as described in Section 5.3.4 1-WEEK FOLLOW-UP OF LENS TYPE #1 (VISIT 3), points 1 to 5.
- 2. Study lens collection at 1-week: investigator will remove study lenses from participant eyes while wearing a pair of disposable non-latex medical grade gloves. The lenses will be rinsed and stored according to sponsor instructions which will be provided at a later date. They will be labeled with study name, participant study ID, eye, visit# and date without any identifying characteristics. They will be stored in a -80 degrees centigrade freezer and shipped to the sponsor when all participants have completed the study.



#### 5.3.7 STUDY EXIT

The study exit form will be completed when a participant exits the study. This form will be completed either at study completion, or if the participant is discontinued from the study at another time. A study exit form must be completed for all participants who have taken a study ID number. If in the opinion of the investigator post-study follow-up visits are required, the exit form will be completed after the last follow-up visit.

After the exit assessments have been completed, the participant and investigator will complete the study completion and remuneration forms. At this time the participant will be considered as having exited the study.

#### 5.3.8 UNSCHEDULED VISITS

An unscheduled visit is defined as an interim visit requested by the participant or investigator due to an unanticipated problem. Data recorded at these visits will be entered into the database. Only relevant and applicable unscheduled visit information will be included in the final report as deemed necessary by the lead investigator.

#### 5.4 STUDY PROCEDURES

The summary of the visits and study procedures to be conducted at scheduled visits is listed in Table 3.

V1 V2 at-home V3 V4 at-home V5 V-Exit Screen Disp ratings 1-week Disp ratings 1-week progress (days progress & fit lens#1 (days lens#2 1,3,5) lens#1 1,3,5) lens#2 lens#1 lens#2 Consent process X CL history and/or lens X X X X X wear schedule Health & medication X X X X X Review any problems with eyes/study lenses X

Table 3: Summary of procedures to be conducted at scheduled visits

| | V1<br>Screen<br>& fit | V2<br>Disp<br>lens#1 | at-home<br>ratings<br>(days<br>1,3, 5)<br>lens#1 | V3<br>1-week<br>progress<br>lens#1 | V4<br>Disp<br>lens#2 | at-home<br>ratings<br>(days<br>1,3, 5)<br>lens#2 | V5<br>1-week<br>progress<br>lens#2 | V-Exit |
|---|---|---|---|---|---|---|---|---|
| Study lens fitting (both lens types) | X | | | | | | | |
| Dispense study CLs* | | X | | | X | | | |
| | x | X | | X | X | | x | |
| Trial lens fit | X | | 9 | | | | | |
| | | X | N. | X | X | | X | |
| Study CL fit assessment | х | Х | | X | X | | X | |
| Complete 'in-office' subjective ratings | | х | 7 | x | x | | х | |
| | | | | | | _ | | |
| | | | | X | | | x | |
| Worn lens collection | | | | X | | | X | |
| | X | X** | // | X | X** | | X | X** |
| Study completion and<br>Exit | | | | | | | | X |

<sup>\*</sup> Additional lenses may be dispensed at scheduled or U/S visits if there is lens defect, or lens damage or if there is a valid reason (e.g. lenses dropped or misplaced etc.)

<sup>&</sup>lt;sup>1</sup>High Contrast High Illumination



#### 6 MONITORING PROTOCOL ADHERENCE

Adherence to study visit windows, lens wearing schedule, and time windows around other data collection points (i.e. subjective ratings) will be monitored internally by CORE. Deviations from the study plan as described in the protocol will be reported in the study report. As described in Section

<sup>\*\*</sup> Not required if visit concurrent with previous one.

15.4, major protocol deviations will be reported to the Sponsor and the University of Waterloo's Office of Research Ethics (ORE) within 7 days of becoming aware of them (as per ORE's guidelines).

#### 7 POTENTIAL RISKS AND BENEFITS TO HUMAN PARTICIPANTS

This is a minimal risk study because of the use of approved products and standard optometric assessments.

Contact lenses in this study will be worn on a daily wear and daily disposable basis. Adverse events and/or complications in the daily wear of soft contact lenses can occur (e.g. inflammation and infection). Complications that may occur during the wearing of contact lenses include discomfort, dryness, aching or itching eyes, excessive tearing, discharge, hyperemia and variable or blurred vision. More serious risks may include photophobia, iritis, corneal edema or eye infection. Although contact lens-related infections are very infrequent, the possibility does exist. The incidence of infection due to daily-wear soft lenses is 0.035%. Almost always an infection will occur only in one eye. Thirty five million Americans who currently wear contact lenses assume this risk.

When contact lenses are worn on a daily wear basis there is a small risk of an adverse event compared to not wearing contact lenses. When contact lenses are worn on an extended wear basis, there is a significantly increased risk of an adverse reaction compared with wearing contact lenses on a daily wear basis.

Additionally, it is possible that participants may experience temporary discomfort associated with the study procedures /products including: burning and stinging, blurred vision, sandiness or grittiness, light sensitivity, dryness, itching, crusty eyes and foreign body sensation.

Participants may not benefit directly from taking part in this study, other than having an opportunity to wear a different contact lens. However, their participation in this study may contribute to scientific research information that may be used in the development of new contact lens products.

Information from this study may help researchers determine new soft contact lens designs to help other people in the future. This study will help the study sponsor to better understand the performance of the products being used in this study.

#### 8 ADVERSE EVENTS

See CORE SOP012\_v02 for a description of all adverse events, including management and reporting. An 'adverse event' refers to any undesirable clinical occurrence in a participant, whether

it is considered to be device-related or not. Adverse events (AE) may be classified as 'unanticipated adverse device effects,' 'serious adverse events,' 'significant adverse events,' or 'non-significant adverse events,' as defined below, Table 4.

A number of conditions may result in temporary suspension until resolution. These include corneal infiltrates, corneal staining, limbal injection, bulbar injection or tarsal conjunctival abnormalities.

Table 4: Classification of types of adverse event

| Classification | Definition |
|---|---|
| Serious Adverse<br>Event | Those events that are life-threatening, or result in permanent impairment of a body function, or permanent damage to a body structure or necessitate medical (therapeutic) or surgical intervention to preclude permanent impairment of a body function or permanent damage to a body structure. |
| Significant<br>Adverse Event | Those non-serious adverse events that occur with contact lens usage that are not sight-threatening but are usually symptomatic and may warrant therapeutic management and /or temporary or permanent discontinuation of contact lens wear. |
| Non-Significant<br>Adverse Events | Those less severe non-serious adverse events that occur with contact lens usage that are not sight-threatening, may or may not be symptomatic and may warrant palliative management, such as ocular lubricants or temporary interruption of contact lens wear. |
| Unanticipated<br>Adverse Device<br>Effect | Adverse events in a study that were not previously identified in the protocol in terms of nature, severity, or degree of incidence. An Unanticipated Serious Adverse Device Effect is an unanticipated adverse event that is serious in nature and caused by or associated with the device and is considered reportable. |

AE classification, coding (for reporting to the sponsor) and reporting details, plus examples, are provided in Table 5.

Table 5: Contact lens adverse event classification, coding and reporting guide

| Code | Condition | Reporting |
|---|---|---|
| Serious Adverse Events | | |
| 01 | Presumed infectious keratitis or infectious corneal ulcer | For all serious |
| 02 | Permanent loss of ≥ 2 lines of best spectacle corrected visual acuity (BSCVA) | AEs: |
| 03 | Corneal injury that results in permanent opacification within central cornea (6mm) | Notify sponsor as soon as possible, |
| 04 | Uveitis or Iritis (e.g. presence of anterior segment inflammation as described in ISO 11980, Annex B) | within 24 hours; |

| 05 | Endophthalmitis | ORE reporting will be within 24 hours as per requirements |
|---|---|---|
| 06 | Hyphema | |
| 07 | Hypopyon | requirements |
| 08 | Neovascularization within the central 6mm of cornea | |
| 00 | Other serious event | |
| Significant Adverse Events | | |
| 11 | Peripheral (outside central 6mm), non-progressive, non-infectious ulcer | |
| 12 | Symptomatic corneal infiltrative event | |
| 13 | Superior epithelial arcuate lesions (SEALs) involving epithelial split | |
| 14 | Corneal staining ≥ dense coalescent staining up to 2mm in diameter (e.g. moderate, ISO 11980 grade 3) | Notify sponsor as soon as possible, within 5 working days; ORE reporting as per requirements |
| 15 | Corneal neovascularization ≥ 1.0mm vessel penetration (e.g. ≥ ISO 111980 Grade 2), if 2 grade change from baseline | |
| 16 | Any temporary loss of ≥ 2 lines BSCVA for ≥ 2wks | |
| 17 | Any sign and/or symptom for which participant is administered therapeutic treatment or which necessitates discontinuation of lens wear for ≥ 2 weeks | |
| 10 | Other significant event | |
| Non-significant Adverse Events | | |
| 21 | Conjunctivitis (bacterial, viral or allergic) | |
| 22 | Papillary conjunctivitis if ≥ mild scattered papillae/follicles approximately 1mm in diameter (e.g. ISO 11890 Grade 2), if 2 grade change from baseline | Notify sponsor as soon as possible, within 5 working days; ORE reporting as per requirements |
| 23 | Asymptomatic corneal infiltrative events | |
| 24 | Any sign and/or symptom for which temporary lens discontinuation for > 1 day is recommended (if not already classified) | |
| 20 | Other sign and/or symptom warranting classification as a non-significant adverse event | |

#### 8.1 NORMAL OR ADAPTIVE SYMPTOMS

Transient symptoms such as end-of-day dryness, lens awareness, itching or burning or other discomfort may occur with contact lens wear and may occasionally reduce wearing time. These are

not reported as adverse events unless in the investigator's opinion they are unexpected in nature, severe or have a high rate of occurrence.

#### 8.2 PROCEDURES FOR ADVERSE EVENTS

Treatment of an adverse event will depend on its nature and severity. Based on the clinical judgment of the investigator the participant may be referred to an ophthalmologist for treatment. The investigator will attempt to determine whether the reaction is related to the test device or a result of other factors. An adverse event form will be completed for each adverse event. If both eyes are involved, a separate adverse event form will be completed for each eye. Whenever possible, the adverse event will be photo-documented.

Expenses incurred for medical treatment as part of study participation will be paid by the sponsor (bills and prescription receipts kept). The participant must be followed until resolution or no further change is anticipated and/or referred for further care with the appropriate health care professional and/or recorded as being under appropriate health care as per investigator's discretion. A written report will be completed indicating the subsequent treatment and resolution of the condition.

#### 8.3 REPORTING ADVERSE EVENTS

All potential Serious and Unanticipated Adverse Device Effects that are related or possibly related to participant's participation will be reported to the Principal Investigator and the sponsor within 24 hours of the investigator becoming aware of the event. The Investigator will report the event to the IRB as per IRB requirements (by fax, mail/delivery, phone, or email). All fatal or life threatening events will be reported immediately to the IRB.

Significant and Non-Significant Adverse Events will be reported to the sponsor as soon as possible, but no later than 5 working days after the occurrence. The Investigator will report the event to the ORE as per ORE requirements (by fax, mail/delivery, phone, or email).



Details of all adverse events will be included in the study report.

#### 9 DISCONTINUATION FROM THE STUDY

Participants discontinued from a study will be reimbursed \$20 per hour for their active involvement in the study (including the initial screening visit). Participants will be discontinued at the discretion of the investigator or sponsor in consideration of participant safety or protocol compliance, or at discretion of the participant. The following is a list of possible reasons for discontinuation from the study:

- Screening failure: Participants will be discontinued if they do not meet the inclusion and exclusion criteria outlined in section 5.1.3.
- Unacceptable performance with products to be used in study: Participants may be discontinued if they are unable to achieve acceptable comfort and /or vision with the study products.
- Positive slit lamp finding: Participants may be permanently discontinued from the study depending on the severity of the condition and on the judgement of the investigator.
- Adverse event: If a participant experiences an adverse event during the study they may be discontinued based on the clinical judgement of the investigator.
- Symptoms: If the participant has persistent symptoms they may be discontinued based on the clinical judgement of the investigator.
- Disinterest, relocation or illness: The participant may choose to discontinue due to reasons within or beyond their control.
- Violation of protocol or non-compliance: The participant will be discontinued if they are unable or unwilling to follow the protocol specified visit schedules and/or study procedures.
- Instillation of topical ocular medication: The participant will be discontinued if they elect to
  use a topical ocular medication during the study unless that topical ocular medication is
  prescribed for a limited duration (less than two weeks) to treat a transient condition; in this
  case the participant may remain an active participant (at the discretion of the investigator)
  after stopping topical ocular medication following resolution of the ocular condition).
- Lost to follow-up: The participant will be discontinued if they cannot be contacted and do
  not return for a final exit visit, and if the investigator has made a reasonable effort to
  contact the participant for a final study visit.
- Premature termination of the study by the sponsor, CORE or the Office of Research Ethics at the University of Waterloo.

A discontinuation form, stating the reason for discontinuation will be completed, which requires the signatures of both the participant and the investigator, except where the participant is lost to follow-up in which case only the signature of the investigator is required.

When a participant choses to discontinue from the study they will be given the opportunity to withdraw their data from the statistical analysis. This choice will be captured on the discontinuation form.

All discontinuations including their reasons will be included in the final report.

#### 10 DEVICE MALFUNCTIONS

A device malfunction means the failure of the device to meet its performance specification or otherwise perform as intended. Any defective lens that is *likely* to cause or contribute to a *Serious Adverse Event* should be reported to the Principal Investigator and the sponsor **within 24 hours** of the investigator becoming aware of the malfunction. The ORE would also be notified within 24 hours of any device malfunction that may contribute to a *Serious Adverse Event*.

Other defective lenses should be reported to the Sponsor as soon as possible (usually in weekly study updates to the Sponsor).

This clinical study will also ascertain satisfaction or preference with subjective attributes such as comfort, vision, or lens handling. Responses to these subjective questionnaires will not be considered as complaints or device malfunctions.

#### 11 STUDY COMPLETION AND REMUNERATION

At the last scheduled protocol visit a study completion form will be completed, which requires the signatures of both the participant and the investigator. Once their involvement in the study is complete, participants will be informed about receiving feedback following study completion in the Letter of Appreciation. Participant remuneration will be \$20 per scheduled protocol visit hour (including the initial screening visit). Full details are given in the information consent letter.

#### 12 STATISTICAL ANALYSIS AND DATA MANAGEMENT

#### 12.1 STATISTICAL ANALYSIS

Primary comparisons will be between study lenses, however there are some variables collected over time with the same lens and this time comparison will be analysed (e.g. 'at-home ratings on Days 1, 3 and 5).

All data will be analyzed by CORE at the University of Waterloo. Unmasked data analysis will be conducted using Statistica, SPSS, or other appropriate software. Descriptive statistics will be provided on information regarding baseline variables (age, gender, refractive error distribution, etc.). Table 6 lists the main outcome variables and anticipated statistical procedures. All data will be tested for normality of distribution using Shapiro-Wilk tests.



Table 6: Statistical analysis to be conducted

| Variable | Analysis | Statistical test |
|---|---|---|
| | Descriptive and other statistics | Mean, Median*, Standard<br>Deviation, Minimum, Maximum,<br>Frequency count |
| Subjective ratings | Effect of treatment on outcome variable within subjects (comparison between study days) Effect of time on ratings (comparison over time) | Friedman<br>Wilcoxon matched pairs test |
| | Descriptive statistics | Mean, Median*, Standard<br>Deviation, Minimum, Maximum,<br>Count |
| | Effect of treatment on outcome variable within subjects (comparison between study days) | RMANOVA<br>Paired t-test |

<sup>\*</sup> For non-parametric data only

The critical alpha level for statistical significance will be set at 0.05, with no adjustments for multiple comparisons.

All participants who were evaluated will be included in the analysis, unless their removal is agreed by the sponsor due to protocol deviations and/or adverse events. In the event of missing data, individual data points will not extrapolated from the collected data.

#### 12.2 DATA MANAGEMENT

Data from this study will be retained by CORE for a minimum of 25 years on a password-protected server. After 25 years, data will be disposed of in accordance with the guidelines laid out by the University of Waterloo.

At the completion of the study CORE will provide a copy of the study data to the sponsor when requested. All data will typically be sent using a secure file share system operated by the University of Waterloo called Sendit which uses 128bit (or 256bit) SSL encryption. This system provides a secure way to transfer files when email is not appropriate, whether because of file size, file type or concerns over security. Sendit includes features such as password protection, a restricted time period for download, IP logging and email notification of download. Files may be encrypted prior to transmission at the request of the sponsor. Using this method means that data files are only stored on University of Waterloo servers until they are downloaded by the sponsor.

#### 12.3 COMMENTS ON SOURCE DOCUMENTS

Data analysis will not be conducted on comments which have been recorded in the source documents, however all comments will be entered into the study database. Only relevant and applicable comments will be included in the final report as deemed necessary by the lead investigator.

#### 13 PROTOCOL TRAINING

All study personnel will be required to complete training prior to their involvement in the study.

#### 14 STUDY MONITORING

Status reports will be provided to the study sponsor by email on a regular basis. Status reports will include:

- The number of participants screened, enrolled, and randomized (i.e. assigned a study ID number), discontinued and completed.
- Details of any protocol deviations.
- Details of any adverse events.

Reports of unintended events.

Study monitoring visits may be conducted throughout the study and will be scheduled by the study sponsor in conjunction with the lead investigator. In addition study records may be inspected at CORE by the sponsor, the sponsor's designate, the Office of Research Ethics at the University of Waterloo, and by regulatory authorities in Canada and the United States, namely Health Canada and the United States Food and Drug Administration (FDA); however, no records containing identifiable/personal information will be permitted to leave the custody of CORE.

#### 15 STUDY MANAGEMENT

#### 15.1 STATEMENT OF COMPLIANCE

This clinical study is designed to be in compliance with the ethical principles in the Declaration of Helsinki, with the ICH guidelines for Good Clinical Practice (GCP), with the University of Waterloo's Guidelines for Research with Human Participants and with the Tri-Council Policy Statement: Ethical Conduct for Research Involving Humans, 2<sup>nd</sup> Edition.

- Declaration of Helsinki
- ICH E6 International Conference on Harmonisation; Good Clinical Practice
- http://iris.uwaterloo.ca/ethics/human/guidelines/index.htm
- http://iris.uwaterloo.ca/ethics/human/ethicsReview/UWStatement.htm
- http://www.pre.ethics.gc.ca/eng/policy-politique/initiatives/tcps2-eptc2/Default/

#### 15.2 ETHICS REVIEW

This protocol will be submitted to and reviewed through the Office of Research Ethics (ORE) at the University of Waterloo. Notification of ethics clearance of the application is required prior to the commencement of the study.

#### 15.3 CLINICAL TRIAL REGISTRATION

This study will be registered with ClinicalTrials.gov by the study sponsor.

#### 15.4 PROTOCOL DEVIATIONS

Protocol deviations are unanticipated or unintentional changes to a study after it has received prior sponsor approval and ethics clearance. Protocol deviations can be major or minor.

#### 15.4.1 MAJOR PROTOCOL DEVIATIONS

Major protocol deviations may impact the research protocol, information consent document or other study materials, usually cannot be anticipated ahead of time and are often necessary to ensure the safety and welfare of the participants.

The following are examples of protocol deviations that must be reported to the ORE:

- Changes in procedures initiated to eliminate immediate risks/hazards to participants;
- Enrollment of participants outside the protocol inclusion/exclusion criteria whether agreed to or not by the sponsor;
- Medication / device / intervention errors (i.e. incorrect drug or dosage of drug / incorrect contact lens(es) dispensed / incorrect care system dispensed);
- Inadvertent deviation in specific research intervention procedures or timing of the research intervention which could impact upon the safety or efficacy of the study-related intervention or upon the experimental design;
- Information consent documentation violations: no documentation of informed consent;
   incorrect version of, or incomplete, informed consent documentation used.

#### 15.4.2 MINOR PROTOCOL DEVIATIONS

Protocol deviations caused by or which originate with research participants are considered minor, and normally are not reported to the ORE unless these result in increased risk to the participant(s). The following are examples of protocol deviations that are considered minor and do not require reporting to the ORE:

- Logistical or administrative aspects of the study (e.g., study participant missed appointment, change in appointment date);
- Inadvertent deviation in specific research intervention procedures or timing of the research intervention which would not impact upon the safety or efficacy of the study-related intervention or upon the experimental design (i.e., missing a measurement during a session that is not considered critical for the study).

#### 15.4.3 REPORTING AND DOCUMENTING PROTOCOL DEVIATIONS

Major protocol deviations must be reported to the ORE within 7 days of the deviation occurring (or its discovery) using the Protocol Deviation Report Form 107 (PDRF). Information from the PDRF is provided to the Clinical Research Ethics Committee (CREC) at the next monthly meeting.

All protocol deviations (major and minor) occurring during the study will be documented and included in the final report.

#### 15.5 PREMATURE TERMINATION OF THE STUDY

The sponsor, CORE or the Office of Research Ethics at the University of Waterloo may terminate the study at any time for any reason.

#### 15.6 STUDY PARTICIPANT RECORDS

Study participant records will be completed to comply with GCP guidelines. Records will contain:

- Unique study acronym and/or code;
- Participant ID;
- Date enrolled;
- Confirmation by investigator that participant met eligibility criteria;
- Confirmation that participant received a signed and dated copy of informed consent;
- Exit date:
- Investigator's signature confirming study exit.

#### 15.7 RETENTION OF STUDY RECORDS AND DATA

Records and data from this study will be retained for a minimum of 25 years. Details regarding storage procedures are given in CORE SOP014 v01 Clinical data management.

#### 16 REPORT

A report will be sent to the sponsors according to terms described in the study contract.

# 1. REFERENCES 1. Section 1. Section 2. Sect